CLINICAL TRIAL: NCT03033173
Title: Ratio of the Cross Sectional Area of Median Nerve to Ulnar Nerve in Diagnosing Carpal Tunnel Syndrome
Status: Completed | Type: Observational
Sponsor: Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: TCRD-TPE-102-05
Record Dates: First submitted 2017-01-18; First posted 2017-01-26 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: An Innovative Diagnostic Method for Carpal Tunnel Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- CTS group
- Healthy subjects

SUMMARY:
An innovative diagnostic ultrasound method for carpal tunnel syndrome was proposed and compared between carpal tunnel syndrome patients and healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* CTS patients were required to have subjective symptoms of numbness, tingling pain, or dysesthesia over the median nerve innervated area of the involved hand.
* Patients should have positive response in either Tinel's test or Phalen's test during physical examination
* Evidence of median neuropathy at wrist level in NCS.
* Control subjects should have neither symptoms nor signs of CTS along with no abnormal findings in electrodiagnostic study of the median nerve and the ulnar nerve across the wrist joint.

Exclusion Criteria:

* Age younger than 20 years old
* Electrodiagnostic evidence of ulnar neuropathy at the wrist level
* Previous trauma or surgery history of hand
* Medical history of hypothyroidism, diabetes mellitus, uremia, rheumatoid arthritis, amyloidosis, and acromegaly
* Pregnancy

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: CTS patients were recruited from the Physical Medicine and Rehabilitation Department of Taipei Tzu Chi hospital.
  Healthy subjects were recruited from hospital staff, health volunteers and their friends.
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Sonographical findings between hands with CTS and healthy hands | Within one week after ultrasound examination

REFERENCES:
- [Derived] Chang YW, Hsieh TC, Tzeng IS, Chiu V, Huang PJ, Horng YS. Ratio and difference of the cross-sectional area of median nerve to ulnar nerve in diagnosing carpal tunnel syndrome: a case control study. BMC Med Imaging. 2019 Jul 4;19(1):52. doi: 10.1186/s12880-019-0351-3. PMID 31272405